CLINICAL TRIAL: NCT04903171
Title: Effects of Enriched Gardens on Cognition and Independence of Nursing Home Residents With Dementia: a Cluster-controlled Trial
Brief Title: Effects of Enriched Gardens in Nursing Home Residents With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RIVAGES (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RIVAGES
Record Dates: First submitted 2021-03-03; First posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer; Enriched garden; Enriched environment; Dementia; Cognitive impairment; Functional autonomy
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Cluster controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigators and outcomes assessor do not know which groups the participants belongs to
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GROUP ONE (No Intervention): The participants do not receive incentive to visit any gardens
- GROUP TWO (Placebo Comparator): The participants receive incentives by carers to visit regularly a conventional sensory garden
  Interventions: Other: INCENTIVE VISITING A GARDEN : ENRICHED OR CONVENTIONAL SENSORY GARDEN
- GROUP THREE (Experimental): The participants receive incentives by carers to visit regularly an enriched garden
  Interventions: Other: INCENTIVE VISITING A GARDEN : ENRICHED OR CONVENTIONAL SENSORY GARDEN

INTERVENTIONS:
Other: INCENTIVE VISITING A GARDEN : ENRICHED OR CONVENTIONAL SENSORY GARDEN — Carers invites every the participants of group 2 and 3 visiting their respective gardens (enriched or conventional sensory garden)
  Arms: GROUP THREE; GROUP TWO

SUMMARY:
Comparing the effect of the frequentation of an enriched garden vs sensory conventional garden by nursing home residents with Alzheimer disease. The effects will be evaluated as regards to cognitive impairment (MMSE), autonomy (ADL) and prevention of falls (Unipodal stance and UpandGo Test)

DETAILED DESCRIPTION:
The cluster controlled trial is conducted over a six months period after recruitment of residents from 4 different nursing homes in France. The participants are distributed into 3 groups. One group does not receive incentive from carers to visit any garden, the second group receives incentives to visit regularly a conventional sensory garden and the third group receive incentives from carers to visit regularly an enriched garden. The study is conducted over a period of 6 months. All participants are giving consent to the study. They will be evaluated before and after over 4 different tests. MMSE (Mini Mental Status Examination) for cognitive impairment, ADL (Activity for day Living) for functional autonomy, TUG (Test up and Go) and Unipodal Stance for prevention of falls.

ELIGIBILITY:
Inclusion Criteria:

* Give consent
* Ability walking alone
* Alzheimer's disease

Exclusion Criteria:

* No dementia
* Severe dementia
* Severe behavioural disorder
* Inability to walk alone

Ages: 75 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 130 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Change in global cognitive function | 6 MONTHS
  Mini Mental Status Examination (MMSE) , 0-30, higher score is the better outcome
Change in functional independence | 6 MONTHS
  Activities of daily living (ADL), 0-6, higher score is the better outcome

SECONDARY OUTCOMES:
Change in gait ability | 6 MONTHS
  Timed Up and Go test (sec), higher time is the worse outcome
Change in balance | 6 MONTHS
  Unipodal Stance (sec), higher time is the better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires Pitié Salpêtrière - Charles Foix et Sorbonne Université, Ivry-sur-Seine, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No
IPD will only be available to study reviewers